CLINICAL TRIAL: NCT02921932
Title: A Randomized Control Trial on the Impact of Prehabilitation Bundle on Perioperative Outcome for Frail Elderly Patients Undergoing Major Abdominal Surgery
Brief Title: The Impact of Prehabilitation Bundle on Perioperative Outcome for Frail Elderly Patients Undergoing Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/2
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Complication, Postoperative; Perioperative/Postoperative Complications
Keywords: Physiotherapy; Inspiratory Muscle Training; Perioperative Medicine; Postoperative outcomes; Preoperative nutrition; Elderly, frail
MeSH Terms: conditions — Postoperative Complications | interventions — Glucerna; Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): In the interventional arm, patients will be given:
  1. A 'Threshold' Inspiratory Muscle Trainer
  2. A nutritional assessment: if needed, dietary supplements prescribed (i.e Ensure, Glucerna).
  3. Cognitive exercise in the form of the 'Memory' card game will be taught to the patients and the caregiver (if available), to be done twice a day.
  Patients will be provided with a protocol activities log and a study assistant will be conducting a telephone conversation on day 1, 4 and 7 to encourage compliance to the protocol and answer any queries with regards to the research study.
  Interventions: Dietary Supplement: Ensure, Resource 2.0 and Glucerna; Other: Cognitive Training, Memory Card Game; Device: 'Threshold' Inspiratory Muscle Trainer, Respironics of New Jersey Inc
- Control (No Intervention): In the control arm, patients will be given the standard education materials regarding surgery and carry out daily activities as usual until the admission of the surgery.

INTERVENTIONS:
Dietary Supplement: Ensure, Resource 2.0 and Glucerna — Preoperative nutritional supplement for undernourished patients
  Arms: Intervention
Other: Cognitive Training, Memory Card Game — Preoperative memory card game
  Arms: Intervention
Device: 'Threshold' Inspiratory Muscle Trainer, Respironics of New Jersey Inc — Inspiratory muscle trainer protocol for strengthening respiratory muscles
  Arms: Intervention

SUMMARY:
This study aims to study the efficacy of a preoperative "bundle" of interventions, which consists of preoperative physiotherapy, nutritional support and cognitive exercises on elderly frail patients undergoing major abdominal surgery, and evaluating their outcomes. There will be two arms, intervention and control.

DETAILED DESCRIPTION:
Frailty is a geriatric syndrome, defined as an increased vulnerability to stressors leading to a state of decreased physiological resistance. It is characterised by a "constellation of symptoms and signs that describe the heterogeneous response of older adults to physiological and metabolic challenges." While frailty is not necessarily synonymous with chronological age, it is more prevalent among the older adult population and is associated with up to a threefold increased risk of mortality or major morbidity postsurgery. Thus, it has become critically important for healthcare systems to develop strategies designed to improve clinical outcomes in this high-risk population when undergoing surgeries.

Currently there is no clear intervention that has been proven to modify the syndrome of frailty or its impact on postoperative outcomes. This study investigates a novel multidisciplinary approach that can be implemented within a short time frame prior to surgery.

We plan to study the efficacy of a preoperative "bundle" of interventions, which consists of preoperative physiotherapy, nutritional support and cognitive exercises on elderly frail patients undergoing major abdominal surgery, and evaluating their outcomes based 1) length of hospital stay 2) Functional recovery from surgery 3) post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients attending the Preoperative Evaluation Clinic, SGH at least 11 days prior to his/her elective major abdominal surgery. Major abdominal surgery is defined as an intraperitoneal surgery with expected length of stay beyond 2 days. For patients who attended the clinic more than 11 days prior to surgery date, they will be informed to start their prehabilitation bundle 10 days prior to surgery.
2. Aged 65 and above
3. Diagnosed as frail based on Fried criteria score 3and above
4. Able to understand and follow the prescribed cognitive and physical exercise

Exclusion Criteria:

1. Patients with Parkinson disease, previous stroke, neuromuscular disorders and those taking carbidopa/levodopa, donepezil hydrochloride or antidepressants as previous studies have found that these medications may cause symptoms that are similar with domains of frailty.
2. Patients who are not able to communicate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay | Will be compared between the intervention and control arms for up to 1 year

SECONDARY OUTCOMES:
Post operative complications | Duration of hospital admission for up to 30 days
  mortality, Intensive Care Unit (ICU) stay, reintubation and ventilation days in ICU, Acute Myocardial Infarction, new arrhythmia.
Functional Post Operative Recovery | Duration of hospital admission for up to 30 days
  Postoperative Quality of Recovery Scale (PQRS) questionnaire at 4 time points (Day of surgery, Postoperative days 1, 3 and 7) throughout their surgical admissions

CONTACTS AND LOCATIONS:
Overall Officials: Hairil R Abdullah, mbbs, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdullah HR, Lien VP, Ong HK, Er PL, Hao Y, Khan SA, Liu CW. Protocol for a single-centre, randomised controlled study of a preoperative rehabilitation bundle in the frail and elderly undergoing abdominal surgery. BMJ Open. 2017 Aug 4;7(8):e016815. doi: 10.1136/bmjopen-2017-016815. PMID 28778994